CLINICAL TRIAL: NCT01555541
Title: A Phase II Study of Intensive Consolidation and Stem Cell Mobilization Therapy With Ofatumumab, Etoposide, and High-dose Ara-C (OVA), Followed by Autologous Stem Cell Transplantation in High-risk Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Brief Title: Intensive Consolidation and Stem Cell Mobilization Therapy Followed by Autologous Stem Cell Transplantation in High-risk Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: C. Babis Andreadis (Other)
Collaborators: University of California, San Francisco (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, C. Babis Andreadis, Assistant Clinical Professor, Department of Medicine, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112525; NCI-2012-00863 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2012-03-09; First posted 2012-03-15 (Estimated); Results first posted 2019-05-17 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Diffuse Large Cell Lymphoma Relapsed/Refractory
Keywords: relapsed; refractory; DLBCL; lymphoma; B-cell; diffuse
MeSH Terms: conditions — Recurrence; Lymphoma | interventions — ofatumumab; Etoposide; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single-arm study (Experimental)
  Interventions: Drug: Ofatumumab; Drug: Etoposide; Drug: Cytarabine

INTERVENTIONS:
Drug: Ofatumumab — 1000 mg IV days 0, 7, 14, 21
  Other Names: Arzerra; GSK1841157; HuMax-CD20
Drug: Etoposide — 10 mg/Kg IV over 24 hours daily, days 1-4
  Other Names: Vespid®; VP-16
Drug: Cytarabine — 2000 mg/m2 IV twice daily, days 1-4
  Other Names: Cytosar-U®; Ara-C; Cytosine arabinoside

SUMMARY:
The goal of this clinical trial is to show that incorporating ofatumumab instead of rituximab in combination with etoposide and cytarabine (OVA) is successful in collecting autologous stem cells for use in an autologous stem cell transplantation (autoSCT) and to examine its effectiveness in eliminating residual diffuse large B-Cell Lymphoma (DLBCL) in patients.

DETAILED DESCRIPTION:
Patients with relapsed Diffuse Large B-cell Lymphoma (DLBCL) who are refractory to or relapse within 12 months of first-line rituximab-based therapy, have poor outcomes with conventional approaches to autologous stem cell transplantation as detailed above. The investigators hypothesize that the intensive mobilization strategy developed can overcome some of the obstacles to successful autologous stem cell transplantation (ASCT) by both eliminating residual disease following salvage therapy and by facilitating stem cell collection. Even though there is clinical experience in the cooperative group setting with intensive pre-ASCT mobilization, it has never been prospectively validated in DLBCL and concerns exist as to its ability to improve outcomes with ASCT in this high-risk, and heavily pretreated group of patients. Furthermore, most patients in the study site's registry treated with intensive mobilization were rituximab-naïve and the findings may not translate in the rituximab-refractory population. The investigators also believe that ofatumumab, a novel monoclonal antibody against a distinct cluster of differentiation antigen 20 (CD20) epitope may in fact overcome rituximab resistance in DLBCL patients and through more effective complement dependent cytotoxicity (CDC) may eliminate minimal residual disease in the patient and contaminating tumor cells in the stem cell graft.

General Design

This is a single-institution, single-arm, prospective phase II study. Patients with high-risk DLBCL (defined as either achieving less than complete remission (CR) to initial rituximab-containing therapy or relapsing within 12 months of initial therapy) will be enrolled on this study and will undergo staging prior to receiving intensive mobilization with ofatumumab, etoposide, and high-dose ara-C (OVA). Following successful stem cell collection, patients will proceed to standard autologous transplantation with cyclophosphamide, 1,3-bis(2-chloroethyl)-1-nitrosourea (BCNU), and etoposide (CBV) preparative regimen. Response evaluation will occur after salvage therapy, following intensive mobilization therapy (d42), at day +90 after ASCT, and at 6, 12 and 24 months thereafter. Event-free, progression-free, and overall survival will also be assessed until 48 months. The primary study endpoint is mobilization-adjusted complete metabolic response rate (maCR) following OVA. Subjects who are not chemosensitive to salvage therapy (i.e. do not achieve a partial response or complete response) will be re-evaluated after an additional salvage regimen. If they are still not chemosensitive at this point, they will be withdrawn from the study and replaced.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of refractory or relapsed biopsy-proven CD20+ diffuse large B-cell lymphoma or primary mediastinal B-cell lymphoma.
* Age 18 years or older
* Refractory to or relapse following a rituximab/anthracycline first-line regimen
* High-risk disease as defined by one of the following:

  * First relapse after CR within 12 months of initiation of front-line therapy
  * Less than CR to front-line therapy
  * Second-line age-adjusted International Prognostic Index score (sAAIPI) of 1 or higher at the time of relapse
* Receipt of no more than three prior chemotherapy regimens. Monoclonal antibody therapy alone and involved field radiotherapy are not included in this number. Prior use of ofatumumab is allowed if there has been no disease progression following that therapy (i.e. ofatumumab-based salvage regimens are allowed)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.

Eligibility to proceed to OVA

* Chemosensitive disease as defined by at least a partial response to salvage therapy by positron emission tomography/computed tomography (PET/CT) criteria.
* Bone marrow with less than 15% lymphoma cells following salvage therapy. No evidence of myelodysplasia.
* Patients must have adequate organ function with serum creatinine <2.0 mg/dL, total bilirubin ≤2 times the upper limit of normal (ULN), and aspartate aminotransferase (AST) ≤3 times the ULN.
* Neutrophils >1,000/μL and platelets >100,000/μL prior to day 0
* No active uncontrolled infection.

Eligibility to proceed to CBV ASCT

* Patients must be out of the hospital after OVA for a minimum of 4 weeks.
* Adequate peripheral blood stem cell collection with cluster of differentiation 34 (CD34) cell dose ≥2 X 106 /kg (actual body weight).
* No evidence of disease progression on day 42 assessment
* Approved by the University of California, San Francisco (UCSF) Bone Marrow Transplant Committee to proceed with ASCT.

Exclusion Criteria

* Presence of disease transformation from a previously diagnosed low-grade lymphoma
* Progression following prior ofatumumab-based therapy
* Active central nervous system or meningeal involvement by lymphoma. Patients with a history of central nervous system (CNS) or meningeal involvement must be in a documented remission by cerebrospinal fluid (CSF) evaluation and contrast MRI imaging for at least 3 months prior to study entry.
* Evidence of myelodysplasia on any bone marrow biopsy.
* Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half-lives or 4 weeks prior to enrollment, whichever is longer, or currently participating in any other interventional clinical study.
* Other past or current malignancy. Subjects who have been free of malignancy for at least 3 years, or have a history of completely resected non-melanoma skin cancer, or successfully treated in situ carcinoma are eligible.
* Chronic or current infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis and active Hepatitis C.
* History of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae
* Known HIV infection
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to randomization, congestive heart failure (NYHA III-IV), and arrhythmia unless controlled by therapy, with the exception of extra systoles or minor conduction abnormalities.
* Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease which in the opinion of the investigator may represent a risk for the patient.
* Positive serology for Hepatitis B (HB) defined as a positive test for HbsAg and a detectable hepatitis B virus (HBV) DNA viral load. If negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HBV DNA test will be performed and if positive the subject will be excluded. If HBV DNA is negative, subject may be included but must undergo at least every 2-month HBV DNA polymerase chain reaction (PCR) testing from the start of treatment during the treatment course. Prophylactic antiviral therapy may be initiated at the discretion of the investigator.
* Positive serology for hepatitis C (HC) defined as a positive test for hepatitis C antibody (HCAb), in which case reflexively perform a hepatitis C virus (HCV) PCR to confirm the result
* Pregnant or lactating women. Women of childbearing potential must have a negative pregnancy test at screening.
* Women of childbearing potential, including women whose last menstrual period was less than one year prior to screening, unable or unwilling to use adequate contraception from study start to one year after the last dose of protocol therapy. Adequate contraception is defined as hormonal birth control, intrauterine device, double barrier method or total abstinence.
* Male subjects unable or unwilling to use adequate contraception methods from study start to one year after the last dose of protocol therapy.
* Subjects who have received live virus vaccination within the 4 weeks prior to planned initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-05-25 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charalambos Andreadis, MD, MSCE, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thiruvengadam SK, Hunter B, Varnavski A, Fakhri B, Kaplan L, Ai WZ, Pampaloni M, Huang CY, Martin T 3rd, Damon L, Andreadis CB. Ofatumumab, Etoposide, and Cytarabine Intensive Mobilization Regimen in Patients with High-risk Relapsed/Refractory Diffuse Large B-Cell Lymphoma Undergoing Autologous Stem Cell Transplantation. Clin Lymphoma Myeloma Leuk. 2021 Apr;21(4):246-256.e2. doi: 10.1016/j.clml.2020.11.005. Epub 2020 Nov 11. PMID 33288485

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: OVA Treatment:
  Ofatumumab: 1000 mg IV days 0, 7, 14, 21
  Etoposide: 10 mg/Kg IV over 24 hours daily, days 1-4
  Cytarabine: 2000 mg/m2 IV twice daily, days 1-4
  ---------
  After Day 42 assessment:
  Autologous Transplantation:
  Stem Cell Infusion on day 0
  Carmustine (BCNU) 15 mg/Kg, day -6
  Etoposide 60 mg/Kg, day -4
  Cyclophosphamide: 100 mg/Kg, day -2
Period: Salvage Response Assessment
Arm/Group | Treatment
Started | 19
Completed | 19
Not Completed | 0
Period: OVA Treatment
Arm/Group | Treatment
Started | 19
Completed | 19
Not Completed | 0
Period: Autologous Stem Cell Transplantation
Arm/Group | Treatment
Started | 12 (7 patients did not move forward due to non-response/progression on last line of therapy prior to Autologous Stem Cell Transplantation (ASCT))
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment: OVA Treatment:
  Ofatumumab: 1000 mg IV days 0, 7, 14, 21
  Etoposide: 10 mg/Kg IV over 24 hours daily, days 1-4
  Cytarabine: 2000 mg/m2 IV twice daily, days 1-4
  ---------
  After Day 42 assessment:
  Autologous Transplantation:
  Stem Cell Infusion on day 0
  BCNU 15 mg/Kg, day -6
  Etoposide 60 mg/Kg, day -4
  Cyclophosphamide: 100 mg/Kg, day -2
Arm/Group | Treatment
Number analyzed (Participants) | 19
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 1
  30-39 years | 1
  40-49 years | 4
  50-59 years | 7
  60-69 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 1
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 19
Cancer Stage at Diagnosis [Count of Participants; unit: Participants] — Stage refers to the extent of the cancer, such as how large the tumor is, and if it has spread. Stages range from 1 (I) to 4 (IV) with higher numbers indicating how larger the cancer tumor is and the more it has spread into nearby tissues.
  Participants
    Stage I - II | 5
    Stage III - IV | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving Complete Response (CR) to the Treatment Upon Successful Stem Cell Mobilization
Description: CR will be calculated based on the PET/CT scan following 2 cycles of salvage therapy using the revised International Working Group (IWG) Criteria for a lymphoma response. This includes: Complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy, Post-treatment residual mass of any size is permitted as long as it is PET-, Spleen and/or liver, if enlarged before therapy based on physical exam or CT scan, should not be palpable on physical exam and should be considered normal size by imaging studies, and nodules related to lymphoma should disappear, If bone marrow was involved by lymphoma before treatment, infiltrate must have cleared on repeat bone marrow biopsy. Biopsy sample must be adequate (with goal of > 20 mm unilateral core). If sample is indeterminate by morphology, it should be negative by immunohistochemistry. A sample that is negative by immunohistochemistry but demonstrates small population of clonal l
Time Frame: Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 19
Participants | 10

2. Primary Outcome: Number of Patients Achieving Mobilization-adjusted Complete Response (maCR)
Description: Number of patients achieving maCR to the treatment upon successful stem cell mobilization, defined as at least 2 x10^6 cluster of differentiation 34 (CD34)+cells/Kg of actual body weight. Patients who require use of plerixafor or an autologous bone marrow harvest are considered mobilization failures and will be treated as non-responders.
Time Frame: Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 19
Participants | 10

3. Secondary Outcome: Number of Patients Who Received OVA and Then Met Criteria to Proceed to ASCT and Achieved a CR/Partial Response (PR) Post-ASCT
Description: Determination of CR or PR must meet the revised International Working Group (IWG) Criteria for lymphoma response
Time Frame: Up to 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 19
Participants | 11

4. Secondary Outcome: Number of Patients Who Advance From Partial Response (PR) to Complete (CR)
Description: Fluorodeoxyglucose-positron emission tomography (FDG-PET) conversion rate was used determined the number of participants who improved following OVA Treatment.
Time Frame: Up to 5 months
Population: 7 Patients were evaluable for PR after salvage
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 7
Participants | 2

5. Secondary Outcome: Number of Participants With Successful Neutrophil Engraftments
Description: Neutrophil engraftment is defined as the first day of 3 consecutive days with absolute neutrophil count of >500 cells/microlitre (uL). Response evaluation will occur at day +90 after ASCT, and at 6, 12 and 24 months thereafter
Time Frame: Up to 24 months after ASCT
Population: Participants who received autologous transplant
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
participants | 12

6. Secondary Outcome: Number of Participants With Successful Platelet Engraftments
Description: Platelet engraftment is defined as the first of three consecutive measurements for which the platelet count was > 20,000/uL, and must be at least 24 hours following the last platelet transfusion. Response evaluation will occur at day +90 after ASCT, and at 6, 12 and 24 months after ASCT
Time Frame: Up to 24 months after ASCT
Population: Participants who received autologous transplant
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
participants | 12

7. Secondary Outcome: Median Time to Progression
Description: Time to progression (TTP) is defined as the time from treatment after OVA until documented lymphoma progression or receipt of anti-lymphoma therapy (except for planned post-ASCT radiotherapy) or death due to lymphoma. Patients are to be censored at the time of last followup or death due to another cause
Time Frame: Up to 48 months
Population: Participants receiving OVA
Measure: Median (Full Range); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 19
months | 13.2 [1.4 to 48]

8. Secondary Outcome: Progression Free Survival Rate
Description: The percentage of participants in the study still alive at time of censoring. The time frame defined as the time from day 0 of OVA treatment until lymphoma progression, receipt of anti-lymphoma therapy (except for planned post-ASCT radiotherapy), or death as a result of any cause. Patients will be censored at the time of median follow-up.
Time Frame: Up to 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 19
percentage of participants | 47 [24 to 67]

9. Secondary Outcome: Overall Survival Rate (OS)
Description: The percentage of participants in the study still alive at time of censoring. The time frame is defined as the time from day 0 of OVA treatment until death as a result of any cause. Patients will be censored at the time of last followup
Time Frame: Up to 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 19
percentage of participants | 59 [33 to 78]

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 3/19
Serious Adverse Events (participants affected / at risk) | 4/19
Other Adverse Events (participants affected / at risk) | 9/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=19)
Anal Pain (Gastrointestinal disorders) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=19)
Platelet count decreased (Investigations) | 9 (12)
Neutrophil count decreased (Investigations) | 8 (11)
White blood cell decreased (Investigations) | 4 (5)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (9)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (2)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (4)
Mucositis oral (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 2 (2)
Lung infection (Infections and infestations) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study closed early due to low accrual

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-01-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT01555541/Prot_SAP_002.pdf
  • Informed Consent Form (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT01555541/ICF_001.pdf